CLINICAL TRIAL: NCT01002456
Title: Beta-Blockers in Heart Failure: Pharmacy-level Intervention Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RRP 09-136; VMS #120 (Other: PBM VAMedSAFE)
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Results first posted 2014-10-15 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
Keywords: Adrenergic beta-Antagonists; Guideline Adherence; Drug Prescriptions; target dose
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Level 1: site-specific information (Other): provide site-specific information on nonadherence
  Interventions: Other: Level 1: (provide site-specifi information)
- Level 2: site-, patient-specific info (Other): provide site- and patient-specific information on nonadherence
  Interventions: Other: Level 2 (Provide site- and patient-specific information)

INTERVENTIONS:
Other: Level 1: (provide site-specifi information) — provide site-specific information on non-adherence to guideline
  Arms: Level 1: site-specific information
Other: Level 2 (Provide site- and patient-specific information) — provide site-specific information on non-adherence to guideline as well as list of patients with non-adherent prescriptions
  Arms: Level 2: site-, patient-specific info

SUMMARY:
The overall objective of the proposed pilot study is to begin evaluation of two methods for promoting adherence to guidelines for beta-blocker therapy in heart failure. The design includes site level baseline measurement, feedback, remeasurement after six months, and randomized (by site) comparison samples. The setting is VA sites, with intervention directed at the pharmacy.

DETAILED DESCRIPTION:
Current evidence-based guidelines in VA recommend one of three beta-blockers (carvedilol, metoprolol succinate, or bisoprolol) that have been shown to reduce mortality in heart failure patients with systolic dysfunction, with recommended target doses. However, Pharmacy Benefits Management (PBM) data indicate that prescribing for beta-blockers in heart failure patients that is not in accordance with guidelines is substantial, both in terms of the agent selected and the dose. Sites will be recruited and randomized to two different intensities of intervention to promote adherence to guidelines.

ELIGIBILITY:
Inclusion Criteria:

* VA sites
* Males and females

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madeline McCarren, PhD MPH, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: provide site-specific information
  Level 1 (Provide site-specific information): provide site-specific information on non-adherence to guideline
- Arm 2: provide site- and patient-specific information
  Level 2 (Provide site- and patient-specific information): provide site-specific information on non-adherence to guideline as well as list of patients with non-adherent prescriptions
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 98 | 122
Completed | 98 | 122
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Level 1: site-specific information provided
- Level 2: site- and patient-specific information provided
- Total: Total of all reporting groups
Arm/Group | Level 1 | Level 2 | Total
Number analyzed (Participants) | 98 | 122 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (11.5) | 71 (11.0) | 71 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 95 | 120 | 215
Region of Enrollment [Number; unit: patients]
  United States | 98 | 122 | 220

OUTCOME MEASURES:

1. Primary Outcome: Rate of Adherence to Guideline Prescription
Description: full adherence to guideline medication and dose
Time Frame: 6 months
Measure: Number; unit: patients
Groups:
- Level 1: provide site-specific information
- Level 2: provide site- and patient-specific information
Arm/Group | Level 1 | Level 2
Number analyzed (Participants) | 98 | 122
patients | 4 | 6
Statistical Analysis 1: Comparison: Level 1 vs Level 2; Test type: Superiority or Other; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.1 to 3.2] — Proportional odds ratio to measure the trend of change in concordance with guideline recommendations, with Arm 1 as the comparator

2. Secondary Outcome: Progress Toward Adherence to Guideline Prescription
Description: either change to a guideline agent or dose increase of a guideline agent
Time Frame: 6 months
Measure: Number; unit: patients
Groups:
- Level 1: Provide Site-specific Information: Level 1: provide site-specific information on nonadherence
- Level 2:Provide Site- and Patient-specific Information: Level 2:provide site- and patient-specific information on nonadherence
Arm/Group | Level 1: Provide Site-specific Information | Level 2:Provide Site- and Patient-specific Information
Number analyzed (Participants) | 98 | 122
patients | 10 | 22

ADVERSE EVENTS:
Groups:
- Level 1: Provide Site-specific Information: Level 1: provide site-specific information on non-adherence
- Level 2: Provide Site- and Patient-specific Information: Level 2: provide site-specific information on non-adherence to guideline as well as list of patients with non-adherent prescriptions
Arm/Group | Level 1: Provide Site-specific Information | Level 2: Provide Site- and Patient-specific Information
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/122
Other Adverse Events (participants affected / at risk) | 0/98 | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes